CLINICAL TRIAL: NCT01197729
Title: OPTAMI (Optimierte Therapie Des Akuten Myokard-Infarktes) - Register
Brief Title: OPTAMI (Optimized Therapy of Acute Myocardial Infarction) - Registry
Acronym: OPTAMI
Status: Completed | Type: Observational
Sponsor: Stiftung Institut fuer Herzinfarktforschung (Other)
Collaborators: Klinikum Nürnberg (Other); University Hospital Muenster (Other); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: OPTAMI
Record Dates: First submitted 2010-09-07; First posted 2010-09-09 (Estimated); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Myocardial Infarction; ST-Elevation Myocardial Infarction; Non-ST-Elevation Myocardial Infarction
Keywords: Myocardial infarction; ST-Elevation myocardial infarction; Non-ST-Elevation myocardial infarction; Register; CARDS
MeSH Terms: conditions — Myocardial Infarction; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- STEMI: (ST-Elevation myocardial infarction)
- NSTEMI: Non-ST-Elevation myocardial infarction

SUMMARY:
OPTAMI documents the characteristics of consecutive patients with acute STEMI and NSTEMI in hospital everyday-life in Germany, their acute and adjuvant medication treatment, events until discharge (e.g. mortality, stroke, re-MI), and their medication for secondary prevention at discharge.

In the follow up-period of one year, information is collected concerning events as mortality, stroke, re-MI, coronary interventions (PCI, CABG) and re-hospitalisation.

The implementation of guideline-adjusted therapy in hospital everyday-life is reviewed. The usefulness of the European standard for data acquisition in cardiology (CARDS = Cardiology Audit and Registration Standards) is evaluated.

ELIGIBILITY:
Inclusion Criteria:

* all patients admitted to hospital with an acute ST-Elevation myocardial infarction or with an acute Non-ST-Elevation myocardial infarction, both not older than 24 h

Exclusion Criteria:

* missing informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 3248 (Actual)
Dates: Start 2005-10; Primary Completion 2009-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Documentation of characteristics from consecutive patients with an acute STEMI or an acute NSTEMI in hospital daily routine in Germany. | 10/01/2005-02/01/2009

SECONDARY OUTCOMES:
Documentation of acute invasive and adjuvant medical therapy of STEMI and NSTEMI in hospital daily routine in Germany | 10/01/2005-02/01/2009
Documentation of hospital mortality and non-fatal cerebrovascular complications (stroke, re-myocardial infarction) | 10/01/2005-02/01/2009
Documentation of medication for secondary prevention at hospital discharge | 10/01/2005-02/01/2009
Documentation of the one-year mortality, the non-fatal cerebrovascular complications (stroke, re-myocardial infarction) as well as of the coronar interventions (PCI, Bypass operation) and hospital admissions during the first year post STEMI or NSTEMI | 10/01/2005-02/01/2009
Verification of the benefits of the European Standards for Data Collection for Cardiology (CARDS = Cardiology Audit and Register Standards) in daily hospital routine. | 10/01/2005-02/01/2009
Verification of the implementation of therapy according to the guidelines for STEMI and NSTEMI patients in daily hospital routine in Germany. | 10/01/2005-02/01/2009

CONTACTS AND LOCATIONS:
Overall Officials: Anselm K Gitt, MD, Study Chair — Stiftung Institut für Herzinfarktforschung; Jochen Senges, MD, Study Chair — Stiftung Institut für Herzinfarktforschung
Locations (2):
- Germany (2):
  - Medizinische Klinik und Poliklinik, Universitätklinikum Münster, Münster
  - Klinikum Nürnberg Süd / Cardiology, Nuremberg